CLINICAL TRIAL: NCT02696512
Title: A Phase 1/2,Open-Label Study to Evaluate the Safety and Efficacy of the International Brain Research Foundation (IBRF) Disorders of Consciousness Advanced Care/MultiModal Care Protocol in Patients With Severe Disorders of Consciousness
Brief Title: A Study of IBRF Disorders of Consciousness Advanced Care/MultiModal Care Protocol in Severe Disorders of Consciousness
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Brain Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBRF-01-10
Record Dates: First submitted 2015-11-19; First posted 2016-03-02 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-08

CONDITIONS: Brain Injury
Keywords: Severe Disorders of Consciousness (SDOC); Coma; Vegetative State; Minimally Conscious State
MeSH Terms: conditions — Brain Injuries; Consciousness Disorders; Coma; Persistent Vegetative State | interventions — Minocycline; Lamotrigine; Flumazenil; Lacteol; Thioctic Acid; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IBRF ACP/MCP Group 1 (Experimental): The Treatment group will be receiving a combination of pharmaceuticals (polypharmacy using FDA-approved products) and nutraceuticals (Nutraceutical supplementation) and median nerve stimulation (MNS)
  Interventions: Drug: Polypharmacy using FDA-approved products; Device: Median Nerve Stimulation (MNS); Dietary Supplement: Nutraceutical Supplementation; Other: Standard of Care
- Standard of Care Group 2 (Other): Standard of Care only
  Interventions: Other: Standard of Care

INTERVENTIONS:
Drug: Polypharmacy using FDA-approved products — Battery of medications provided through a 12-week schedule including: Minocycline, Lamotrigine, Flumazenil, Modafinil, Bromocriptine, Donepezil, Methylphenidate, Methyl B12, Methylfolate, Rasagiline, Amantadine, Naltrexone and Levodopa/carbidopa.
  Other Names: Minocycline, Lamotrigine, Flumazenil, and others
  Arms: IBRF ACP/MCP Group 1
Device: Median Nerve Stimulation (MNS) — 40 cycle/second (gamma range) asymmetric, 2 ms wavebands with 300 µs bursts at 20 milliamps bilaterally (randomized left arm and right arm sequencing algorithm) applied 20 seconds on and 40 seconds off for 8 hours per day.
  Other Names: Empi PV300 TENS
  Arms: IBRF ACP/MCP Group 1
Dietary Supplement: Nutraceutical Supplementation — Battery of nutraceuticals provided through a 12-week schedule including: Acidophilus, Alpha-Lipoic Acid, Acetyl L-Carnitine,
  Other Names: Acidophilus, Alpha-Lipoic Acid, and others
  Arms: IBRF ACP/MCP Group 1
Other: Standard of Care — Standard of Care treatment

SUMMARY:
This is a study to evaluate the safety and efficacy of the IBRF ACP/MCP intervention protocol in patients with severe disorders of consciousness (SDOC).

DETAILED DESCRIPTION:
Currently, there are no empirically validated, evidence-based pharmacological interventions for the treatment of Severe Disorders of Consciousness (SDOC). In addition, it is unclear why poly-pharmacological interventions, while more common in the treatment of other disorders (e.g., cancer, chronic pain), have not been embraced for the treatment SDOC; some of the lone agents used in treatment of SDOC patients are not "indicated" for combined treatment.

In addition, the treatment of SDOC traditionally employs the use of single or small combinations of pharmacological agents, with no single pharmacological agent being identified as efficacious or effective. As such, a poly-pharmacological intervention may, inherently, involve pharmacological interactions that were not anticipated by the drug manufacturers or prescribing physicians.

The purpose of this study is to document the safety of the IBRF ACP/MCP and to establish its efficacy for those SDOC patients successfully completing treatment. The IBRF ACP/MCP employs a poly-pharmacological approach aimed at studying arousal states and outcomes in SDOC patients beyond those rates documented in literature.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years to ≤ 65 years
* GCS rating of 3 to 9 (severe impairment)
* Evidence of an acquired brain injury that severely suppresses consciousness
* Coma, vegetative state, or minimally conscious state based on definitions of the Mohonk Report
* If polytrauma, patient is medically stable

Exclusion Criteria:

* GCS of 10 or greater (moderate to mild impairment)
* Tracheostomies requiring ventilator support
* Medical condition that precludes objective assessment (e.g., concurrent Guillain-Barre or other severe peripheral neuropathy, severe critical illness myopathy/polyneuropathy)
* Onset of injury greater than 12 months post hypoxic ischemic injury (HII)
* Onset of injury greater than 24 months post traumatic brain injury (TBI)
* Emergence during the screening period
* Terminal illnesses, existing severe neuro-developmental disorders, existing chronic degenerative neurological conditions, prior moderate-to-severe TBI, or any stroke syndrome other than transient ischemic attack (TIA), or a prior seizure disorder
* Patients with an uncontrolled seizure disorder, or seizure disorder can only be controlled with medication that is contra-indicated (e.g., dilantin or phenobarbitol),
* In the opinion of the attending physician, the patient presents with a cardiac condition that would place them at unacceptable risk, or has a documented ejection fraction (EF) <25%

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-03 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Tolerance to treatment | Week 12
  The percent of patients completing the treatment protocol
Number and Frequency of side effects | Week 12
  The total number and frequency of side effects experienced by patients based on observations and evaluations of the patients' clinical laboratory tests
Adverse events | Week 12
  Based on observations of the study patients and evaluations of clinical laboratory tests

SECONDARY OUTCOMES:
coma recovery scale-revised (CRS-R) | Week 12
disability rating scale (DRS) | Week 12
functional assessment measure (FIM) | Week 12
Glasgow coma scal (GCS) | Week 12
Glasgow outcome scale-extended (GOS-E) | Week 12
orientation log (O-LOG) | Week 12
vegetative state (VS) | Week 12
  Clinical diagnosis (, minimally conscious state; MCS, emerged) using criteria from the Mohonk Reports
minimally conscious state (MCS) | Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Philip A Defina, Ph.D., Principal Investigator — IBRF
Locations (1):
- International Brain Research Foundation, Edison, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes